CLINICAL TRIAL: NCT04979715
Title: The Effect of Early Rehabilitation After Breast Cancer Surgery on Physical and Psychosocial Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, ATİYE KAŞ ÖZDEMİR, Principal Investigator; Phd. PT, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019SABE028
Record Dates: First submitted 2021-06-24; First posted 2021-07-28 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer Surgery
Keywords: breast cancer; physical functions; psychosocial functions; breast cancer physiotherapy; breast cancer survival; breast cancer surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: intervention (Group 1), control (Group 2) and routine follow-up (Group 3) groups
Who Masked: Participant
Masking Description: participants do not know which group they belong to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (Group 1) (Experimental): From the first postoperative day, with the approval of the surgeon performing the operation, the postoperative exercise program will be started once a day under the supervision of a physiotherapist during the stay of the participants in the hospital.
  At the same time, participants will be directed to moderate intensity aerobic exercise (walking, jogging…) for 150 min/week. Information will be given on the importance of physical activity and increasing the level of physical activity. In addition, a brochure containing explanatory information about the postoperative physiotherapy program after breast surgery will be given to the participants.
  Interventions: Procedure: physitherapy follow-up
- control group (Group 2) (Active Comparator): The patients in the control group will be informed about the postoperative physiotherapy program and patient education will be provided by the physiotherapist before the operation. Within the knowledge and approval of the surgeon performing the operation, preoperatively, respiratory control, diaphragmatic breathing, relaxation exercises, passive-active assistive-active range of motion exercises are shown by the physiotherapist, and patient education is provided with information about possible postoperative complications and what needs to be considered. will be given.
  Interventions: Other: control
- routine follow-up (Group 3) (No Intervention): only preoperative patient information is given.

INTERVENTIONS:
Procedure: physitherapy follow-up — preoperative patient informaiton, information leaflet and Physiotherapy meeting will be held every 2 weeks for 3 months
  Arms: intervention group (Group 1)
Other: control — no intervention; preoperative patient informaiton and information leaflet
  Arms: control group (Group 2)

SUMMARY:
At least 42 patients between the ages of 30-65, who were followed up in Pamukkale University General Surgery Breast Polyclinic and planned for breast surgery, will be included in the study. Those who met the criteria for inclusion in the study and those who voluntarily agreed to participate in the study, who were preoperatively evaluated, will be randomly divided into two groups using the closed envelope method by matching age, gender, type of surgery and breast cancer stage. The first of these groups is the study (n=21) and the second is the control group (n=21).

DETAILED DESCRIPTION:
Study group: Patients in the study group will be informed about the postoperative physiotherapy program and patient education will be provided by the physiotherapist before the operation. After obtaining the consent of the surgeon performing the operation, preoperative and post-operative complications (infection, lymphedema, fatigue…) and the things to be considered (use of upper extremities, skin care, importance of weight control…) and patient education will be given by the physiotherapist. In addition, respiratory control, diaphragmatic breathing, relaxation exercises, gradual passive-active assistive-active range of motion exercises, stretching exercises will also be demonstrated preoperatively.

From the first postoperative day, with the approval of the surgeon performing the operation, the postoperative exercise program will be started once a day under the supervision of a physiotherapist during the stay of the participants in the hospital.

At the same time, participants will be directed to moderate intensity aerobic exercise (walking, jogging…) for 150 min/week. Information will be given on the importance of physical activity and increasing the level of physical activity. In addition, a brochure containing explanatory information about the postoperative physiotherapy program after breast surgery will be given to the participants.

Participants will continue the exercises as a home program after discharge. During this follow-up period, the participants will meet again with the physiotherapist every two weeks for the control, compliance and continuity of the exercises. In these interviews, while compliance with the exercise program is checked, exercise tolerance will also be determined and necessary interventions and modifications will be made. In case of any complication (limitation in physical functions, lymphedema…) during the home program, he will be informed about meeting with the relevant physician and physiotherapist as soon as possible.

Control group: The patients in the control group will be informed about the postoperative physiotherapy program and patient education will be provided by the physiotherapist before the operation. Within the knowledge and approval of the surgeon performing the operation, preoperatively, respiratory control, diaphragmatic breathing, relaxation exercises, passive-active assistive-active range of motion exercises are shown by the physiotherapist, and patient education is provided with information about possible postoperative complications and what needs to be considered. will be given.

Written consent of all participants was obtained; demographic information will be recorded, and their physical and psychosocial conditions will be evaluated. Circumference measurements for lymphedema The extremity volume will be calculated using the Frustum formula. Modified Constant Murley Score for shoulder and upper extremity loss of function and evaluation of activities of daily living, pectoralis major and pectoralis minor shortness tests, Tanita for body composition determination, L-Dex score for bioimpedance analysis, Functional Evaluation of Breast Cancer Treatment for functional status ( Functional Assessment of Cancer Therapy -Breast Cancer - FACT-B scale, Cancer Fatigue Scale for fatigue, 6 Minute Walk Test (6MWT) for cardiovascular endurance and Hospital Anxiety and Depression Scale (HAD) for psychosocial status will be used. All measurements will be repeated preoperatively (at least 3 days before the operation), on the 1st postoperative day and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Having a breast surgery indication with a diagnosis of breast cancer
* Having stage 1-2-3 breast cancer
* Education level to be at least literate
* To be in stable clinical condition
* Not having any other disease that will affect their physical and psychosocial functions
* Being good at cooperation
* Referred by the relevant surgeon and no contraindications for early postoperative physiotherapy

Exclusion Criteria:

* History of previous breast cancer surgery
* Concurrent bilateral breast cancer and/or surgery
* History of shoulder surgery
* Preoperative shoulder dysfunction
* Upper extremity deep vein thrombosis
* BMI>40 kg/m²
* Use of an assistive walking device
* Stage 4 metastatic cancer
* All conditions that require close monitoring during exercise (such as uncontrolled or unstable cardiovascular disease or diabetes)
* cognitive impairment

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
determination of limb volume changes | postoperative to 3 months later
  The circumference measurements for lymphedema will be calculated using the Frustum formula. calculations will compare with operated and non-operated limb, and also subsequent measurements. A volume increase of >200 ml is interpreted as the onset of lymphedema.
determination of shoulder and upper extremity functions | postoperative to 3 months later
  Modified Constant Murley Score for assessment of shoulder and upper extremity functions. high score indicates good function.
muscle shortness test | postoperative to 3 months later
  Pectoralis major and pectoralis minor muscle shortness tests.measurements will compare with operated and non-operated limb, and also subsequent.
Bioimpedance analysis for body composition determination; weight | postoperative to 3 months later
  Tanita bioimpedance analysis device will be used to determine body composition. Measurements will be compared with the subsequent. bioimpedance analysis determines that; body weight (kg), muscle mass (kg), estimated bone ratio (kg).
Bioimpedance analysis for body composition determination;body mass index | postoperative to 3 months later
  Tanita bioimpedance analysis device will be used to determine body composition. Measurements will be compared with the subsequent. bioimpedance analysis determines that; body mass index (kg/m2).
Bioimpedance analysis for body composition determination; body fat and water percentage | postoperative to 3 months later
  Tanita bioimpedance analysis device will be used to determine body composition. Measurements will be compared with the subsequent. bioimpedance analysis determines that; body fat percentage, body water percentage.
Bioimpedance analysis for body composition determination; visceral fat level | postoperative to 3 months later
  Tanita bioimpedance analysis device will be used to determine body composition. Measurements will be compared with the subsequent. bioimpedance analysis determines that; visceral fat level.
Bioimpedance analysis for body composition determination; energy consumption | postoperative to 3 months later
  Tanita bioimpedance analysis device will be used to determine body composition. Measurements will be compared with the subsequent. bioimpedance analysis determines that; total daily energy consumption (kcal/day).
Bioimpedance analysis for body composition determination; metabolic age | postoperative to 3 months later
  Tanita bioimpedance analysis device will be used to determine body composition. Measurements will be compared with the subsequent. bioimpedance analysis determines that; metabolic age (years).
determination of subdermal fluid ratio | postoperative to 3 months later
  Moisturemeter compactD for measurement of subdermal fluid ratio. Measurements will be compared with the subsequent.
assesment of fatigue | postoperative to 3 months later
  Cancer Fatigue Scale for assesment of fatigue. A low score indicates a low fatigue rate.
determination of cardiovascular endurance | postoperative to 3 months later
  6 Minute Walk Test (6MWT) will be used for cardiovascular endurance.Changes of >35 m are significant changes.

SECONDARY OUTCOMES:
determination of emotional status | baseline to 3 months later
  It is expected that the psychosocial functions that have decreased due to breast cancer will be restored in a short time with physiotherapy follow-up and improvement of physical functions. Hospital Anxiety and Depression Scale (HAD) will be used for psychosocial status. A low score indicates low anxiety and depression.
Determination of quality of life | postoperative to 3 months later
  Functional Assessment of Cancer Therapy -Breast Cancer (FACT-B) scale for assessment of functional status and activities of daily living. high score indicates good function.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda YILMAZ, dr, Study Chair — Pamukkale University; Hande ŞENOL, dr, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kas Ozdemi̇r A, Telli Atalay O, Yilmaz S, Senol H. The effects of early rehabilitation on physical and psychosocial functions after breast cancer surgery. Support Care Cancer. 2025 Sep 23;33(10):872. doi: 10.1007/s00520-025-09926-4. PMID 40987957